CLINICAL TRIAL: NCT01993563
Title: The Effect of a Graded Motor Imagery Approach for Stroke Patients Within a Year After Stroke
Brief Title: Graded Motor Imagery for Patients Within a Year After Stroke.
Acronym: GMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Principal Investigator, Andrea Polli, MSc, IRCCS San Camillo, Venezia, Italy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GMI_RCT_STROKE
Record Dates: First submitted 2013-11-13; First posted 2013-11-25 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-04

CONDITIONS: Stroke
Keywords: Stroke; Rehabilitation; Motor Imagery; Upper Extremity; Mirror Therapy
MeSH Terms: conditions — Stroke | interventions — Neurological Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Graded Motor Imagery (Experimental)
  Interventions: Other: Graded Motor Imagery
- Standard treatment (Active Comparator)
  Interventions: Other: Standard treatment

INTERVENTIONS:
Other: Graded Motor Imagery — GMI program includes three steps: Implicit Motor Imagery (IMI); Explicit Motor Imagery (EMI) and Mirror Box Therapy (MT).
  IMI included a training based on Hand Laterality Discrimination Tasks. During these tasks 60 pictures of right and left hands are projected randomly on a 15" screen. Patients are asked to choose whether the images seen are right or left and therefore to click respectively the right or the left button on a mouse.
  EMI training consists in imagining a movement without actual performing it. It will be introduced during IMI's last two sessions and gradually enhanced increasing the complexity of motor skills to be imagined. The therapist shows or explains in details the movements the patient have to mentally rehearsed.
  MT treatments will start with simply watching the unaffected hand in the mirror and increased toward functional movement. When possible, gentle movement with the affected hand will be encouraged behind the reflecting part of the mirror.
  Other Names: GMI
  Arms: Graded Motor Imagery
Other: Standard treatment — Patients will undergo to a standard treatment, that is thought to be the best option for that specific patients. In our hospital, treatment options include: motor training, functional training, occupational therapy, bilateral arm training or motor treatment using virtual reality devices.
  Other Names: motor training; neurorehabilitation
  Arms: Standard treatment

SUMMARY:
The aim of the study is to evaluate whether a graded rehabilitation approach including Implicit and explicit motor imagery training and mirror therapy is more effective than other treatments commonly provided in a neuro-rehabilitation department.

DETAILED DESCRIPTION:
Graded Motor Imagery is a graded approach recently proposed for treating chronic pain patients. It included three subsequent steps:

1. Implicit Motor Imagery training (IMI), using a body part laterality discrimination task
2. Explicit Motor Imagery training, using pictures and videos for improving patient's ability in imagining movements
3. Mirror box therapy, using a 35x40 cm mirror,

We are transferring this approach into stroke rehabilitation in order to improve patients' upper limb motor functions.

All the patients, in both groups, will be training 2 hours a day, 5 days/week for 4 weeks. The first hour is standard treatment, the clinician in charge will decide treatment's priorities and the aim(s) of the treatment for each specific patient. The second hour will be focused on patient's upper limb function.

The treatment group will be treated accordingly to the GMI protocol. The control group will receive a second hour of standard treatment, centred on the upper limb. Standard treatments are decided by the interdisciplinary team and might include motor rehabilitation, bilateral arm training, virtual reality training or occupational therapy.

ELIGIBILITY:
Inclusion Criteria:

1. ischemic or hemorrhagic stroke within a year from the event;
2. age of participant between 21 and 85 years old;
3. absence of apraxia or global aphasia;
4. Mini-Mental State Examination score >23.

Exclusion Criteria:

1. Presence of other neurological or orthopaedic disorders affecting upper extremity motor function,
2. Neglect,
3. Significant spasticity defined as a score ≥ 24 total points at Tardieu Rating Scale (TRS)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-10 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change in Wolf's Motor Function Test (WMFT) | before and after the 4-weeks treatment
  It includes 17 different tasks, which assess shoulder, elbow, wrist function and manual ability. For each task, a qualitative mark is given and time needed to complete the action is recorded.
Change in Fugl Meyer Assessment Scale for upper extremity (FMA) | Before and after the 4-weeks treatment
  We use the Upper Extremity session of the scale. The scale evaluates patient's balance, passive and active movements of shoulder, elbow, wrist and hand. It also evaluates different types of grips. Sense of position and ability to detect light touches are also evaluated.

SECONDARY OUTCOMES:
Change in Functional Independence Measure (FIM) | before and after the 4-weeks treatment
  FIM is an 18-item scale developed to assess severity of patient disability and medical rehabilitation functional outcome
Change in Transcranial Magnetic Stimulation (TMS) | before and after the 4-weeks treatment
  In order to assess a possible neurophysiological effect of our treatment, we also evaluate cortical excitability using Single Stimulus TMS.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Turolla, MSc, Study Director — IRCCS Ospedale San Camillo
Locations (1):
- IRCCS Ospedale San Camillo, Venice, Italy, Italy